CLINICAL TRIAL: NCT00289757
Title: Double-blind, Randomized Study to Evaluate the Immunogenicity and Reactogenicity of Three Different Lots of GlaxoSmithKline Biologicals' Inactivated Hepatitis A Vaccine Containing 1440 EL.U of Antigen Per mL and Injected According to a 0, 6 Month Schedule in Healthy Adult Subjects
Brief Title: Long-Term Immune Persistence of GlaxoSmithKline Biologicals' Inactivated Hepatitis A Vaccine, Injected According to 0, 6-month Schedule
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 100576 (Y11); 100577 (Y12) (Other: GSK); 100578 (Y13) (Other: GSK); 100579 (Y14) (Other: GSK); 100580 (Y15) (Other: GSK); 111028 (Y16) (Other: GSK); 111029 (Y17) (Other: GSK); 111030 (Y18) (Other: GSK); 111031 (Y19) (Other: GSK); 111032 (Y20) (Other: GSK)
Record Dates: First submitted 2006-02-09; First posted 2006-02-10 (Estimated); Results first posted 2010-03-04 (Estimated); Last update posted 2018-07-23 (Actual); Status verified 2016-09

CONDITIONS: Hepatitis A
Keywords: Havrix™; Hepatitis A
MeSH Terms: conditions — Hepatitis A | interventions — Hepatitis A Vaccines

ARMS (1):
- Havrix Group (Experimental): Subjects who received 2 doses of Havrix™ (lot A, B or C) in the primary study.
  As lot to lot consistency was assessed during the primary study, the 3 groups (lot A, B or C) were pooled into the Havrix Group for data analyses during the long term follow-up.
  Interventions: Biological: Havrix™

INTERVENTIONS:
Biological: Havrix™ — 2 doses at 6 months interval

SUMMARY:
The aim of this study is to evaluate the long-term persistence of hepatitis A antibodies at 11, 12, 13, 14, 15, 16, 17, 18, 19 and 20 years after subjects received their first dose of a 2 dose vaccination schedule of hepatitis A vaccine.

DETAILED DESCRIPTION:
This is a long-term follow-up study at Years 11, 12, 13, 14, 15, 16, 17, 18, 19 and 20 after primary vaccination with GSK Biologicals' hepatitis A vaccine (two-dose schedule). To evaluate the long-term antibody persistence, volunteers will donate a blood sample at Years 11, 12, 13, 14,15, 16, 17, 18, 19 and 20 after the first vaccine dose of the primary vaccination course to determine their anti-hepatitis A (anti-HAV) antibody concentrations If a subject has become seronegative for anti-HAV antibodies during any of the long-term blood sampling time point (i.e. Years 11, 12, 13, 14, 15, 16, 17, 18, 19 and 20 years), he/ she will be offered an additional vaccine dose. A blood sample will be taken on the day of the additional vaccination, 14 days and one month after additional vaccination to evaluate the immune response following this vaccination.

The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007 and to include an extended follow up period up to Year 20 after primary vaccination.

The study has 10 phases (100576, 100577, 100578, 100579, 100580, 111028, 111029, 111030, 111031, 111032).

ELIGIBILITY:
Inclusion Criteria:

* Subjects who had received at least one dose of the study vaccine in the primary study
* Written informed consent will have been obtained from the subjects before the blood sampling visit of each year.

Ages: 29 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2004-01-01; Primary Completion 2013-03-01 (Actual); Study Completion 2013-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Wilrijk, Belgium

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Desombere I et al. (2000) Long-term persistence of cellular immunity towards hepatitis A vaccine (HAV) following HAV vaccination. J Antiviral Therapy. 5: 7.
- [Background] Van Damme P, Mathei C, Thoelen S, Meheus A, Safary A, Andre FE. Single dose inactivated hepatitis A vaccine: rationale and clinical assessment of the safety and immunogenicity. J Med Virol. 1994 Dec;44(4):435-41. doi: 10.1002/jmv.1890440422. PMID 7897376
- [Background] Van Damme P et al. (1998) Long-term immunogenicity of a high potency inactivated hepatitis A vaccine. J Hepatol. 28 (suppl.1): 113.
- [Background] Van Herck K et al. (2000) Model-based estimates of long-term persistence of vaccine-induced hepatitis A antibodies. J Antiviral Therapy. 5:3-4.
- [Background] Van Herck K, Van Damme P. Inactivated hepatitis A vaccine-induced antibodies: follow-up and estimates of long-term persistence. J Med Virol. 2001 Jan;63(1):1-7. PMID 11130881
- [Background] Van Herck K, Jacquet JM, Van Damme P. Antibody persistence and immune memory in healthy adults following vaccination with a two-dose inactivated hepatitis A vaccine: long-term follow-up at 15 years. J Med Virol. 2011 Nov;83(11):1885-91. doi: 10.1002/jmv.22200. Epub 2011 Aug 23. PMID 21915861
- [Background] Van Herck K, Crasta PD, Messier M, Hardt K, Van Damme P. Seventeen-year antibody persistence in adults primed with two doses of an inactivated hepatitis A vaccine. Hum Vaccin Immunother. 2012 Mar;8(3):323-7. doi: 10.4161/hv.18617. Epub 2012 Feb 13. PMID 22327499
- [Derived] Agrawal A, Kolhapure S, Andani A, Ota MOC, Badur S, Karkada N, Mitra M. Long-Term Persistence of Antibody Response with Two Doses of Inactivated Hepatitis A Vaccine in Children. Infect Dis Ther. 2020 Dec;9(4):785-796. doi: 10.1007/s40121-020-00311-8. Epub 2020 Jul 24. PMID 32710245
- [Derived] Theeten H, Van Herck K, Van Der Meeren O, Crasta P, Van Damme P, Hens N. Long-term antibody persistence after vaccination with a 2-dose Havrix (inactivated hepatitis A vaccine): 20 years of observed data, and long-term model-based predictions. Vaccine. 2015 Oct 13;33(42):5723-5727. doi: 10.1016/j.vaccine.2015.07.008. Epub 2015 Jul 16. PMID 26190091
- [Derived] Hens N, Habteab Ghebretinsae A, Hardt K, Van Damme P, Van Herck K. Model based estimates of long-term persistence of inactivated hepatitis A vaccine-induced antibodies in adults. Vaccine. 2014 Mar 14;32(13):1507-13. doi: 10.1016/j.vaccine.2013.10.088. Epub 2014 Feb 7. PMID 24508042
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 100576 (Y11) — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 100576 (Y11) — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 100576 (Y11) — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 100576 (Y11) — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register. The results of this study 100576 are summarised with studies 100577, 100578, 100579, 100580, 111028, 111029, 111030, 111031, and 111032 on the GSK Clinical Study
- Available data/document: Dataset Specification: 100576 (Y11) — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 100576 (Y11) — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participant Flow and Baseline measures are given for the Month 192 (Year 16) time point in order to account for all subjects participating in this long-term follow-up study. Note that not all subjects returned and participated in each of the intermediate follow-up time points.
Pre-assignment Details: The Long-Term (LT) Total Cohort included all subjects who returned for the follow-up and who belonged to the Total Cohort in the primary study.The Long Term According-to-Protocol (LT-ATP) cohort for immunogenicity included subjects who returned for the follow-up and who were included in the ATP cohort for immunogenicity of the primary study.
Period: Overall Study
Arm/Group | Havrix Group
Started | 78
Completed | 78
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Havrix Group
Number analyzed (Participants) | 78
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.3 (7.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56
  Male | 22

OUTCOME MEASURES:

1. Primary Outcome: Anti-hepatitis A Virus (Anti-HAV) Antibody Concentration
Description: Concentrations given as geometric mean concentration (GMC) expressed as milli-international unit per millilitre (mIU/mL).
  The laboratory assay was changed at Year 11, thus the blood samples were with both the old and the new assay for the sake of bridging.
Time Frame: At Years 11, 12, 13, 14, 15, 16, 17, 18, 19 and 20 after the first vaccine dose of the 2-dose primary vaccination
Population: Analysis was performed on the Long Term According-to-Protocol (LT-ATP) cohort for immunogenicity, on subjects with available data for the defined timepoint.
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Havrix Group
Number analyzed (Participants) | 53
mIU/mL
  Year 11 Old Assay Method (N=43) | 593.6 [452.0 to 779.5]
  Year 11 New Assay Method (N=46) | 297.4 [220.1 to 401.8]
  Year 12 (N=42) | 363.2 [263.1 to 501.2]
  Year 13 (N=50) | 287.7 [218.6 to 378.6]
  Year 14 (N=46) | 270.4 [196.5 to 372.1]
  Year 15 (N=41) | 290.3 [210.7 to 400.1]
  Year 16 (N=53) | 242.3 [182.8 to 321.3]
  Year 17 (N=45) | 277.9 [206.5 to 374.0]
  Year 18 (N=37) | 301.7 [211.2 to 431.1]
  Year 19 (N=26) | 226.5 [154.8 to 331.3]
  Year 20 (N=34) | 311.8 [233.2 to 416.8]

2. Primary Outcome: Anti-hepatitis A Virus (Anti-HAV) Antibody Concentration
Description: Concentrations given as GMC expressed as mIU/mL.
Time Frame: Before the additional dose, 14 days and 30 days after the additional dose
Population: Analysis was performed on the Long Term Total cohort, only on subjects who received an additional vaccine dose during the current long-term follow-up study. If a subject became seronegative (< 15 mIU/mL) at any of the long-term blood sampling timepoint, he/she was offered an additional vaccine dose.
Measure: Number; unit: mIU/mL
Arm/Group | Havrix Group
Number analyzed (Participants) | 2
mIU/mL
  Subject 1 (pre-additional dose) | 23
  Subject 1 (14 days post-additional dose) | 702
  Subject 1 (30 days post-additional dose) | 836
  Subject 2 (pre-additional dose) | 24
  Subject 2 (14 days post-additional dose) | 6107
  Subject 2 (30 days post-additional dose) | 5939

3. Primary Outcome: Number of Seropositive Subjects for Anti-HAV Antibodies.
Description: Seropositivity for anti-HAV antibodies defined as antibody concentrations ≥ 15 mIU/mL for Year 11 to Year 20 time points.
  The laboratory assay was changed at Year 11, thus the blood samples were with both the old and the new assay for the sake of bridging.
Time Frame: From Year 11 to Year 20
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Havrix Group
Number analyzed (Participants) | 53
Subjects
  Year 11 Old Assay Method (N=43) | 43
  Year 11 New Assay Method (N=46) | 46
  Year 12 (N=42) | 42
  Year 13 (N=50) | 50
  Year 14 (N=46) | 46
  Year 15 (N=41) | 41
  Year 16 (N=53) | 53
  Year 17 (N=45) | 45
  Year 18 (N=37) | 37
  Year 19 (N=26) | 26
  Year 20 (N=34) | 34

4. Secondary Outcome: Number of Subjects Reporting Serious Adverse Events (SAE) Assessed by the Investigators as Related to Vaccination or to Study Procedures or Lack of Efficacy
Description: An SAE is any untoward medical occurrence that: results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect in the offspring of a study subject, or may evolve into one of the outcomes listed above
Time Frame: Years 11, 12, 13, 14, 15, 16, 17, 18, 19 and 20 after the first vaccine dose of the 2-dose primary vaccination
Population: Analysis was performed on the Long Term Total cohort which included all subjects who returned to the follow-up study and who had received at least 1 dose of the vaccine in the primary study.
Measure: Number; unit: Subjects
Arm/Group | Havrix Group
Number analyzed (Participants) | 78
Subjects
  Year 11 (N=64) | 0
  Year 12 (N=60) | 0
  Year 13 (N=71) | 0
  Year 14 (N=66) | 0
  Year 15 (N=63) | 0
  Year 16 (N=78) | 0
  Year 17 (N=63) | 0
  Year 18 (N=52) | 0
  Year 19 (N=45) | 0
  Year 20 (N=50) | 0

5. Secondary Outcome: Number of Subjects Reporting Any and Grade 3 Solicited Local Symptoms
Description: Solicited local symptoms assessed include pain, redness and swelling. Grade 3 pain = symptom that prevented normal activities. Grade 3 redness and swelling = redness or swelling above 30 mm and persisting more than 24 hours.
  Any = incidence of a particular symptom regardless of intensity.
Time Frame: During the 4-day (Day 0-3) follow-up period after additional vaccination
Population: as for outcome 2
Measure: Number; unit: Subjects
Arm/Group | Havrix Group
Number analyzed (Participants) | 2
Subjects
  Any Pain | 1
  Any Redness | 0
  Any Swelling | 0
  Grade 3 Pain | 0
  Grade 3 Redness > 30 mm | 0
  Grade 3 Swelling > 30 mm | 0

6. Secondary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Solicited General Symptoms
Description: Solicited general symptoms assessed included fatigue, fever, gastrointestinal symptoms, and headache.
Time Frame: During the 4-day (Day 0-3) follow-up period after additional vaccination
Population: as for outcome 2
Measure: Number; unit: Subjects
Arm/Group | Havrix Group
Number analyzed (Participants) | 2
Subjects
  Any, Grade 3 and Related Fatigue | 0
  Any, Grade 3 and Related Fever | 0
  Any, Grade 3 and Related Gastrointestinal | 0
  Any, Grade 3 and Related Headache | 0

7. Secondary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Unsolicited Adverse Events (AE)
Description: An AE is any untoward medical occurrence in a clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Grade AE = produced significant impairment of functioning or incapacitation and was a definite hazard to the subject's health.
  Related AE = assessed by the investigator as related to the study vaccination.
Time Frame: During the 30-day follow-up period after additional vaccination (for subjects who received the additional vaccine dose between Year 11 and 15)
Population: as for outcome 2
Measure: Number; unit: Subjects
Arm/Group | Havrix Group
Number analyzed (Participants) | 2
Subjects
  Any AE(s) | 1
  Grade 3 AE(s) | 0
  AE(s) Related | 0

8. Secondary Outcome: Number of Subjects Reporting Serious Adverse Events (SAE)
Description: as for outcome 4
Time Frame: During the follow-up period after additional vaccination up to Year 20
Population: as for outcome 2
Measure: Number; unit: Subjects
Arm/Group | Havrix Group
Number analyzed (Participants) | 2
Subjects | 0

ADVERSE EVENTS:
Time Frame: Until year 20 for SAEs and within 4-days after additional vaccination for other AEs. During the 30-day (Day 0 to Day 29) follow-up period after additional vaccination.
Description: Analyses were performed on the Long-Term (LT) Total Cohort including subjects who returned for the follow-up and who belonged to the Total Cohort in the primary study. For the other AEs only subjects receiving an additional dose were included. Therefore the number of subjects at risk is not consistent with the LT Total Cohort.
Arm/Group | Havrix Group
Serious Adverse Events (participants affected / at risk) | 0/78
Other Adverse Events (participants affected / at risk) | 2/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Havrix Group (N=2)
Pain (General disorders) | 1 — Within 4-day period after additional vaccination.
Influenza like illness (Infections and infestations) | 1 — During the 30-day follow-up period after additional vaccination

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.